CLINICAL TRIAL: NCT00596739
Title: Weight Loss Surgery and Male Fertility
Brief Title: A Study of the Pre- and Post-operative Semen Analyses and Reproductive Hormone Levels of Men Undergoing Weight-reduction Surgery
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 805770
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Male Infertility
Keywords: Bariatric surgery, weight loss surgery, male infertility, Roux-En-Y, gastric banding
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Sperm
Oversight: Data Monitoring Committee: No

SUMMARY:
A correlation between obesity and male fertility has been observed in a few clinical studies. Normal weight men appear to have higher sperm concentrations and sperm motility when compared to obese men, suggesting that weight loss might improve sperm function. However, there also are reported cases of severe male factor infertility following weight loss surgery in previously fertile men. The aim of this study is to determine if there are differences in the semen analyses and hormone levels of men obtained before and after undergoing weight loss (bariatric) surgery.

This will direct future research and treatment.

DETAILED DESCRIPTION:
We will recruit 60 subjects for this study. Volunteers will provide pre-operative semen and blood samples prior to undergoing weight-reduction surgery.

Those with normal pre-operative sperm samples will be invited to continue participating in the study by providing subsequent post-operative semen samples and hormonal testing over a two year time period.

It is estimated to take approximately one year to enroll the desired 60 subjects. The study will conclude two years from the last enrollment.

The main analysis will be a comparison of sperm concentrations over time.

ELIGIBILITY:
Inclusion Criteria:

* Adult male subjects between the ages of 18-65 undergoing bariatric surgery

Exclusion Criteria:

* Subjects with abnormal sperm analysis

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male subjects between the ages of 18-65 undergoing bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Changes in semen analyses and reproductive hormone measurements | 2 years

SECONDARY OUTCOMES:
Trends in semen analysis & reproductive hormone parameters over the two-year data collection period, Changes in semen analysis & reproductive hormone parameters as a function of BMI | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Samantha F Butts, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States